CLINICAL TRIAL: NCT05578235
Title: Optimising Surgical Anastomosis in Ileocolic Resection for Crohn's Disease to Reduce Recurrent Disease: A Randomised Controlled Trial Comparing Hand-sewn (END-TO-END or Kono-S) to Stapled Anastomosis (END-to-END Study)
Brief Title: Comparing Hand-sewn (END-TO-END or Kono-S) to Stapled Anastomosis in Ileocolic Resection for Crohn's Disease
Acronym: END2END
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA) (Other)
Collaborators: ZonMw: The Netherlands Organisation for Health Research and Development (Other)
Responsible Party: Principal Investigator, Willem A. Bemelman, Prof. dr., Amsterdam UMC, location AMC
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2022.0533; NL81981.018.22 (Other: CCMO)
Record Dates: First submitted 2022-10-01; First posted 2022-10-13 (Actual); Last update posted 2023-12-18 (Actual); Status verified 2023-11

CONDITIONS: Crohn Disease
Keywords: Crohn's disease; Ileocolic; Endoscopic Recurrence; Ileocolic Anastomosis
MeSH Terms: conditions — Crohn Disease

STUDY DESIGN:
Intervention Model Description: Randomised controlled trial. Patients with Crohn's disease will be randomised in a 1:2 ratio for stapled side-to-side anastomose versus handsewn anastomosis (either end-to-end or Kono-S) when performing an ileocolic resection for Crohn's disease.
Who Masked: Participant, Outcomes Assessor
Masking Description: There is no blinding to the treatment allocation for the treating surgeon. The treatment will be blinded for the treating gastroenterologist, the endoscopist and the participants.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- stapled side-to-side anastomosis (Active Comparator): Standard procedure for CD, ileocolic resection with side-to-side anastomosis is done according to local practice with a linear stapler either aniso- or isoperistaltic as advised by the ECCO guidelines
  Interventions: Procedure: stapled side-to-side anastomosis
- Handsewn anastomosis: handsewn end-to-end or Kono-s anastomosis (Active Comparator): * Kono-S (anti-mesenteric functionel end-to-end handsewn) anastomosis is done according to the description by Kono
  * End-to-end handsewen anastomosis is fashioned either by enlarging the small bowel diameter by an antimesenteric incision to fit the large bowel lumen or by tailored resection of a part of the staple line of the cross stapled colon
  Interventions: Procedure: Handsewn anastomosis

INTERVENTIONS:
Procedure: stapled side-to-side anastomosis — Standard procedure for CD
  Arms: stapled side-to-side anastomosis
Procedure: Handsewn anastomosis — handsewn end-to-end or Kono-s anastomosis
  Arms: Handsewn anastomosis: handsewn end-to-end or Kono-s anastomosis

SUMMARY:
The aim of this multicenter randomised controlled trial is to compare the handsewn (end-to-end and Kono-S) to the stapled side-to-side ileocolic anastomosis after ileocolic resection for Crohn's disease with respect to 6 months endoscopic recurrence, functional outcome and health care consumption.

DETAILED DESCRIPTION:
Within the surgical IBD society there has been a lot of attention to technical aspects of ileocolic resection aiming to reduce recurrent Crohn's disease after surgery. Despite optimal surgical and medical management, recurrent disease after surgery is common. Different types of anastomoses with respect to configuration and construction can be made after resection e.g., handsewn (end-to-end and Kono-S) and stapled (side-to-side). The various types of anastomoses might affect endoscopic recurrence and its assessment, the functional outcome, and costs. It is hypothesised that patients who had an end to end reconstruction will have less endoscopic recurrence (less overscoring, and less stases), a better function and consequently health care consumption than the stapled side to side anastomosis.

ELIGIBILITY:
Inclusion Criteria:

* Males and females aged >16 years
* Ileocolic disease or disease of the neoterminal ileum with an indication for resection
* Concurrent therapies with corticosteroids, 5-ASA drugs, thiopurines, MTX, antibiotics, and anti-TNF therapy are permitted.
* All patients should have undergone a colonoscopy and a recent update of imaging (e.g. Ultrasound, MR enterography (or CT enterography if MR is contraindicated))- Ability to comply with protocol.
* Competent and able to provide written informed consent.
* Patient must have been discussed in the local MDT

Exclusion Criteria:

* Inability to give informed consent.
* Patients less than 16 years of age.
* Clinically significant medical conditions within the six months before the operation : e.g. myocardial infarction, active angina, congestive heart failure or other conditions that would, in the opinion of the investigators, compromise the safety of the patient.
* History of cancer < 5 years which might influence patients prognosis
* Emergent operation.
* Pregnant or breast feeding.
* Inability to follow up at 3, 6 and 12 months for postoperative assessment, imaging and endoscopy.

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 165 (Estimated)
Dates: Start 2023-07-13 (Actual); Primary Completion 2027-10-01 (Estimated); Study Completion 2027-10-01 (Estimated)

PRIMARY OUTCOMES:
Postoperative endoscopic recurrence at 6 months | 6 months
  The postoperative endoscopic recurrence at 6 months following ileocolic resection defined as Rutgeerts > i2b by central reading

SECONDARY OUTCOMES:
Post-operative 30 days complications | 30 days after surgery
Histologic and clinical recurrence rate at 6 months following ileocolic resection | 6 months after surgery
Number of patients in need for restarting immunosuppressive medication within the first year postoperatively for endoscopic or clinical recurrence | 1 year after surgery
  * Endoscopic recurrence defined as Rutgeerts > i2b
  * Clinical recurrence difned as recurrent CD-related symptoms
The 5 year reoperation rate for recurrence of disease at the anastomotic site. | 5 year
Inflammatory Bowel Disease Questionnaire (IBDQ) | 1 year after surgery
  Quality of life measured with IBD questionnaire
Hospital costs | 1 year after surgery
  Hospital costs per patients in each group

CONTACTS AND LOCATIONS:
Overall Officials: W.A. Bemelman, Prof. dr., Principal Investigator — Amsterdam UMC, location AMC
Locations (1):
- Flevoziekenhuis, Almere Stad, Flevoland, Netherlands

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Haanappel AEG, Bellato V, Buskens CJ, Armuzzi A, van der Bilt JDW, de Boer NKH, Danese S, van der Does de Willebois EML, Duijvestein M, van der Horst D, Pellino G, Richir MC, Selvaggi F, Spinelli A, Vignali A, Rosati R, Bemelman WA. Optimising surgical anastomosis in ileocolic resection for Crohn's disease with respect to recurrence and functionality: two international parallel randomized controlled trials comparing handsewn (END-to-end or Kono-S) to stapled anastomosis (HAND2END and the End2End STUDIES). BMC Surg. 2024 Feb 26;24(1):71. doi: 10.1186/s12893-024-02340-3. PMID 38408943